CLINICAL TRIAL: NCT05757596
Title: A Phase 1 Clinical Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Effects of a Single Dose of VSA001 Injection in Chinese Healthy Adult Volunteers
Brief Title: Study of VSA001 Injection in Chinese Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Visirna Therapeutics HK Limited (Industry)
Collaborators: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: VSA001-1001
Record Dates: First submitted 2023-02-14; First posted 2023-03-07 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Healthy Adult Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- VSA001 injection (Active Comparator): A single dose of active drug (VSA001, low or high dose) will be administered by subcutaneous injection on Day 1.
  Interventions: Drug: VSA001 injection
- Placebo (Placebo Comparator): The placebo is normal saline (0.9%) administered subcutaneously; volume matched to the corresponding VSA001 dose volume.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VSA001 injection — The active drug is VSA001 injection. The active pharmaceutical ingredient (API) contained in VSA001 is a synthetic, double-stranded, hepatocyte targeted NAG-conjugated RNAi.
  Arms: VSA001 injection
Drug: Placebo — 0.9% Saline, volume matched
  Arms: Placebo

SUMMARY:
This is a phase 1, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics effects of a single dose of VSA001 injection in Chinese healthy adult volunteers. Eligible enrolled participants will initially receive VSA001 injection at the assigned dose level.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily participate in this study who are able to read, understand, and sign the ICF before participation; and have a full understanding of the content, process and possible adverse reactions of the study and are able to complete the study in accordance with the requirements of the protocol.
2. Healthy male and female subjects aged between 18 and 55 years (both inclusive) at the time of informed consent.
3. Body mass index (BMI) = weight (kg)/height (m)2, within the range of 19.0-30.0 kg/m2 (both inclusive), and body weight no less than 50 kg.
4. In good general health and without clinically significant abnormalities as judged by the investigator, based on medical history, physical examination, vital signs, 12-lead ECG, and laboratory results.
5. Negative serum pregnancy test within 72 h prior to initiation of study treatment in all premenopausal females and females who have been amenorrheic for less than 12 months. (Serum pregnancy test is not required for females who have undergone surgical sterilization, such as hysterectomy and/or bilateral oophorectomy, or those who have not experienced menses for 12 consecutive months and are judged to be postmenopausal based on factors such as age and castration therapy).
6. Subjects and their partners must agree to use adequate contraceptive methods prior to initiation of study treatment, during the study, and for at least 3 months after discontinuation of study treatment.
7. Fasting serum TGs >80 mg/dL (>0.903 mmol/L) at screening.

Exclusion Criteria:

1. History or presence of significant or clinically significant diseases/abnormality, including but not limited to cardiac/cardiovascular, respiratory, endocrine, gastrointestinal, renal, hepatic, gallbladder, dermatological, hematological, immunological, neurologic, or psychiatric diseases/abnormality, or the disease that, in the judgement of the investigator, present a safety concern or affects the pharmacokinetic evaluation.
2. A family history of congenital long QT syndrome, Brugada syndrome or unexplained sudden cardiac death.
3. Subjects who are with acute exacerbation of any significant acute or chronic disease as judged by the investigator.
4. AST and ALT >2×upper limit of normal (ULN) , or total bilirubin >ULN at screening.
5. Serum creatinine estimated eGFR < 60 ml/min/1.73 m2 per MDRD formula.
6. Cardiac troponin (troponin I) above ULN at Screening.
7. Fasting serum TGs >300 mg/dL (>3.38 mmol/L) at screening.
8. Presence of other conditions or treatments that may affect the study results and interfere with the subject's participation in the study as assessed by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 85 days
  Incidence, frequency, and severity of adverse events (AEs) and serious adverse events (SAEs), and the relationship with VSA-01001.
  Clinically significant abnormalities in laboratory tests, vital signs, physical examination, 12-lead electrocardiograms (ECG).

SECONDARY OUTCOMES:
Pharmacokinetics parameter: Cmax | 48 hours
  Maximum plasma concentration (Cmax)
Pharmacokinetics parameter: Tmax | 48 hours
  Time to maximum plasma concentration (Tmax)
Pharmacokinetics parameter: AUC0-t | 48 hours
  Area under the plasma concentration-time curve from the time 0 to the last quantifiable time point (AUC0-t).
Pharmacokinetics parameter: t1/2 | 48 hours
  Half-life (t1/2).
Pharmacokinetics parameter: CL/F | 48 hours
  Apparent clearance (CL/F).
Pharmacokinetics parameter: Vz/F | 48 hours
  Apparent volume of distribution (Vz/F).
Pharmacodynamic (PD) parameters | 85 days
  Change from baseline over time in fasting serum APOC3 and triglycerides (TGs).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang F, You D, Niu X, Shi J, Li Y, Qi L, Li H. Safety, pharmacokinetics and pharmacodynamics of Plozasiran in Chinese healthy volunteers. Cardiovasc Diabetol. 2025 Oct 15;24(1):399. doi: 10.1186/s12933-025-02929-9. PMID 41094680